CLINICAL TRIAL: NCT02382445
Title: Anesthesia Depth Increases the Degree of Postoperative Dementia, Delirium, and Cognitive Dysfunction by a Higher Load of Neurotrophic Drugs
Brief Title: Anesthesia Depth Increases the Degree of Postoperative Dementia, Delirium, and Cognitive Dysfunction
Acronym: BIS & Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Thomas Frietsch, Prof. Dr. med. Thomas Frietsch, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIS-Diako-Ma-2014
Record Dates: First submitted 2014-08-11; First posted 2015-03-06 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia; Delirium; Dementia; Bispectral Index Monitor
MeSH Terms: conditions — Delirium; Dementia | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anesthesia depth monitor (Experimental): Anesthesia depth is aimed to be between BIS 50-60
  Interventions: Device: Anesthesia depth monitor; Drug: propofol and sevoflurane
- Control group (Sham Comparator): Anesthesia depth is monitored but blinded to the anesthesiologist
  Interventions: Device: Sham control; Drug: propofol and sevoflurane

INTERVENTIONS:
Device: Anesthesia depth monitor
  Other Names: Aim at an anesthesia level of BIS 50-60 titrating propofol and sevoflurane in the experimental
  Arms: Anesthesia depth monitor
Device: Sham control — Standard care as usual. Bis m Standard care as usual. Bispectral index monitor is not visible for anesthesia provider.
  Arms: Control group
Drug: propofol and sevoflurane

SUMMARY:
Anesthetics and anesthesia are suspicious to induce dementia or aggravate preexistent cognitive deficits with or without evoking postoperative delirium. In animal trials various anesthetics induce increased levels of misfolded amyloid beta and protein tau, the molecular substance of pathophysiologic brain tissues of demented patients. The amount of those markers seems to correlate well with the degree of dementia [1]. In contradiction, a single study indicates that the incidence of postoperative cognitive deficit (POCD) decreases if hypnotic depth is deep [2]. Unfortunately the study did not sum up the amount of anesthetic drug load, since this would have clarified if the amount of anesthetics used is associated to POCD and dementia. Another possibility is that stress and noxious stimulation induced by light anesthesia results in POCD, whereas deep anesthesia protects from it or inhibits implicit memory.

The investigators' prospective randomized trial is underway to verify the impact of anesthetics and narcotic depth upon grade of dementia and incidence of early postoperative cognitive dysfunction on postoperative day 1 as well as the incidence of delirium within a 90 day period.

The investigators' hypothesis is that the incidence of POCD and delirium and the degree of early cognitive dysfunction is less when anesthetic and vasoactive drug load is less in the BIS- guided anesthesia group with the superficial but sufficient anesthesia level.

ELIGIBILITY:
Inclusion Criteria:

* adults older than 70 years
* major surgery ( spine, orthopedic, urologic, gynecology, abdominal)

Exclusion Criteria:

* adults younger than 71 years
* major blood loss surgery
* allergy to soja oil, nuts, other ingredients of propofol
* patient wants to have spinal or regional anesthesia only

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-01; Primary Completion 2017-05-08 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Postoperative cognition and mental capacity of elderlies following major surgery | One day after surgery
  Mini Mental State Test (MMSE) and automated Memory and Attention Test (MAT) were performed on the day before and after the surgery. The MAT is a validated computerized test for the discrimination of short and long time memory, for visual and auditory comprehension and attention capacity.

SECONDARY OUTCOMES:
Incidence of mental and other complications (serious adverse events) | 90 postoperative days
  Incidences of delirium and mental dysfunction until hospital discharge is counted. Delirium was postoperatively diagnosed by the NUDESC, postoperative cognitive dysfunction (POCD) by the MAT, other serious adverse events in the course of the hospital stay were noted.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frietsch, Prof, MD, Study Director — Universitätsmedizin Mannheim
Locations (1):
- Diakonissen Hospital, Mannheim, Baden-Wurttemberg, Germany